CLINICAL TRIAL: NCT06878521
Title: Strengthening Emotional Regulation: a Preliminary Efficacy Study of a Group Intervention with Adolescents [Fortaleciendo La Regulación Emocional: Un Estudio De Eficacia Inicial De Una Intervención Grupal Con Adolescentes]
Brief Title: Strengthening Emotional Regulation: a Group Intervention with Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lorena Wenger Amengual (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Sponsor-Investigator, Lorena Wenger Amengual, Principal Investigator, Universidad de La Frontera
Organization: Universidad de La Frontera (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FONDECYT INI 11230147
Record Dates: First submitted 2025-01-29; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-01

CONDITIONS: Emotional Regulation
Keywords: Adolescents; Emotional regulation; Transdiagnostic; Transdiagnostic intervention; Group intervention; Emotion Regulation Skills Training; School-based intervention
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial (RCT) with a parallel-group design and a waitlist control group. Participants will be randomly assigned to one of two groups:
  1. Experimental Group: This group will receive the emotional regulation skills training (ERST) intervention immediately.
  2. Control Group: This group will not receive the intervention initially but will be placed on a waitlist and receive the same ERST intervention after the experimental group has completed the program.
  This design allows for a direct comparison between the experimental and control groups during the initial intervention period, ensuring that any observed effects can be attributed to the ERST program. The waitlist control group ensures that all participants eventually receive the intervention, maintaining ethical standards.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emotional regulation skills training Group (Experimental): Participants in this group will receive the emotional regulation skills training (ERST) intervention.
  Interventions: Other: Emotional Regulation Skills
- Waitlist Control Group (No Intervention): Participants in this group will not receive the intervention initially and will be placed on a waitlist. They will receive the same emotional regulation skills training (ERST) intervention after the experimental group has completed the program.

INTERVENTIONS:
Other: Emotional Regulation Skills — This intervention is inspired by and incorporates elements of Dialectical Behavior Therapy (DBT). It consists of eight weekly group sessions, each lasting approximately 1.5 to 2 hours, held on school premises. Each group includes 8 to 10 adolescents. The sessions are facilitated by two psychologists and/or senior psychology students who have been specifically trained to deliver the intervention.
  The sessions focus on developing various emotional regulation skills, which participants are encouraged to practice both during and between sessions. Some of the key skills covered include Mindfulness, Wise Mind, and Problem-Solving, among others.
  Arms: Emotional regulation skills training Group

SUMMARY:
The goal of this clinical trial is to determine the initial efficacy of an emotional regulation skills training (ERST) intervention program in a group of adolescents presenting mild symptoms affecting their ability to regulate emotions. For this purpose, a sample of 1st and 2nd-year high school students (ages 14-16) will be recruited, and the intervention will be conducted on the educational institution's premises during school hours. The main questions it aims to answer are:

Does the ERST intervention reduce symptom levels in adolescents with mild emotional dysregulation? Does the ERST intervention improve emotional regulation skills in adolescents? Researchers will compare pre-intervention (T1) and post-intervention (T2) outcomes, as well as follow-up assessments at 3 months, to evaluate changes in symptom levels and emotional dysregulation. Additionally, a blinded teacher assessment will be conducted at T1 and T2 to evaluate symptom levels.

Participants will:

Attend the ERST intervention sessions during school hours. Complete self-report assessments at four time points (T1, T2, and 3-month follow-up).

Be evaluated by a blinded teacher at T1 and T2.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents in their first or second year of high school.
* Must be currently enrolled in school.
* They should be referred for emotional dysregulation issues and require mental health support.
* They must score above the 75th percentile on the total scale of the SDQ screening tool

Exclusion Criteria:

* Adolescents who are regularly receiving psychological treatment

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Emotional Dysregulation Over Time Compared to the Control Group | Day 0 = during enrollment, Month 2 = immediately after the experimental group completes the intervention, and Month 3 = three months later for follow-up
  Emotional dysregulation is measured using the "Difficulty in Emotion Regulation Scale" (DERS-E). This self-report questionnaire is administered to participants at baseline (Day 0), at the end of the intervention (Month 2), and three months later for follow-up (Month 3).
Change from Baseline in Psychological Functioning screening Over Time Compared to the Control Group | Day 0 = during enrollment, Month 2 = immediately after the experimental group completes the intervention, and Month 3 = three months later for follow-up
  Psychological functioning screening is assessed using the "Strengths and Difficulties Questionnaire" (SDQ) (self-report version), which measures emotional and behavioral difficulties. The minimum value for the general difficulty scale is 0, and the maximum value is 40, where higher scores indicate worse psychological functioning.
  This questionnaire is administered to participants at baseline (Day 0), at the end of the intervention (Month 2), and three months later for follow-up (Month 3).
Change from Baseline in Anxiety Symptoms Over Time Compared to the Control Group | Day 0 = during enrollment, Month 2 = immediately after the experimental group completes the intervention, and Month 3 = three months later for follow-up
  Anxiety Symptoms are assessed using the "Generalized Anxiety Disorder 7" (GAD-7), which measures the presence and severity of anxiety symptoms. The minimum value for the scale is 0, and the maximum value is 21, where higher scores indicate worse anxiety symptoms.
  This questionnaires is administered to participants at baseline (Day 0), at the end of the intervention (Month 2), and three months later for follow-up (Month 3).
Change from Baseline in Depressive Symptoms Over Time Compared to the Control Group | Day 0 = during enrollment, Month 2 = immediately after the experimental group completes the intervention, and Month 3 = three months later for follow-up
  The evaluates the severity of depressive symptoms.
  Depressive Symptoms are assessed using the "Patient Health Questionnaire 9" (PHQ-9), which measures the severity of depressive symptoms. The minimum value for the scale is 0, and the maximum value is 27, where higher scores indicate worse depressive symptoms.
  This questionnaires is administered to participants at baseline (Day 0), at the end of the intervention (Month 2), and three months later for follow-up (Month 3).

SECONDARY OUTCOMES:
Change from Baseline in Clinical Symptoms Over Time Compared to the Control Group, with Masking in the Evaluation Process | Day 0 = during enrollment, Month 2 = immediately after the experimental group completes the intervention
  A blinded teacher assessment will be conducted at baseline (Day 0), at the end of the intervention (Month 2) to evaluate symptom levels in both groups, using the "Strengths and Difficulties Questionnaire: Teacher-rated" (SDQ). The minimum value for the general difficulty scale is 0, and the maximum value is 40, where higher scores indicate worse psychological functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de La Frontera, Temuco, Chile